CLINICAL TRIAL: NCT01801202
Title: Clinical Evaluation of LightSheer Duet 805nm HS Handpiece
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Lumenis Be Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: LUM-ABU-HS 805nm-12-01
Record Dates: First submitted 2013-02-21; First posted 2013-02-28 (Estimated); Last update posted 2015-04-29 (Estimated); Status verified 2014-08

CONDITIONS: Hair Removal

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hair removal (Experimental): hair removal treatment using 805nm LightSheer Duet HS handpiece
  Interventions: Device: LightSheer Duet HS handpiece

INTERVENTIONS:
Device: LightSheer Duet HS handpiece — The approach to be studied here relies on a cleared modality, the LightSheer Duet High Speed (HS) that uses 805 nm diode laser with vacuum (K053628).

SUMMARY:
* The study will re-confirm that the LightSheer Duet HS 805 nm handpiece is safe for removal of unwanted hair, and will result in hair removal and permanent hair count reduction.
* Twenty (20)subjects, Fitzpatrick Skin Type I-IV will be included in a single site.
* Each subject will receive five treatments at four to six week intervals and return for follow-up visits at three and six months after the last treatment for evaluation of the treated areas.

ELIGIBILITY:
Inclusion Criteria:

1. Able to read, understand and provide written Informed Consent;
2. Healthy adult, male or female, 18 years of age or older with skin type I-IV;
3. Having a suitable treatment area for hair removal;
4. Able and willing to comply with the treatment/follow-up schedule and requirements;
5. Women of child-bearing potential (women who have not had a hysterectomy, bilateral oophorectomy or are not postmenopausal) are required to be using a reliable method of birth control at least three months prior to enrollment and throughout the course of the study.

Exclusion Criteria:

1. Pregnant, expectation of pregnancy, postpartum or nursing (<6 months);
2. Hormonal disorders that may affect hair growth;
3. Immunosuppressive diseases, including AIDS and HIV infection, or use of immunosuppressive medications;
4. Livedo reticularis;
5. Uncontrolled systemic diseases such as diabetes;
6. Active infections in the treated area;
7. Dysplastic nevi;
8. Significant concurrent skin conditions or any inflammatory skin conditions;
9. Active cold sores, open lacerations or abrasions;
10. Chronic or cutaneous viral, fungal, or bacterial diseases;
11. Current cancer;
12. History of skin cancer or pre-cancerous lesions at the treatment areas;
13. Use of Accutane™ (Isotretinoin) within the past six month;
14. Keloid formation in the treatment area;
15. Tattoos in the treatment area;
16. Bleeding coagulopathies or use of anticoagulants;
17. Auto-immune disorders;
18. Erythema ab igne, when identified treatments should be discontinued;
19. Photosensitivity disorder that can be exacerbated by laser or intense light;
20. Herpes simplex in the treatment area;
21. Use of medications, herbal supplements, perfumes or cosmetics that may affect sensitivity to light;
22. Poor wound healing;
23. Sunburns;
24. Unable or unlikely to refrain from artificial tanning, including the use of tanning booths, prior (at least a week) and during the course of the evaluation;
25. Prior skin treatment with laser or other devices on the same treated areas within the last six months prior to study enrollment or during the course of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2013-02; Primary Completion 2014-11 (Actual); Study Completion 2014-11 (Actual)

PRIMARY OUTCOMES:
Number of subjects with Adverse Events | 1 year
  To evaluate the safety of hair removal using the LightSheer Duet HS 805 nm handpiece
Hair count | 6 monts follow up
  To verify hair removal and permanent hair reduction using the LightSheer Duet HS 805 nm handpiece

SECONDARY OUTCOMES:
Subject's comfort using VAS | Baseline, 4, 8, 12, 16 weeks;
  To evaluate subject's assessment of comfort associated with treatments
Asses subject's perception of improvement and satisfaction | 8, 16 weeks following baseline; 3 and 6 monts follow up
  To evaluate subject's satisfaction with hair removal treatments and assessment of improvement using subject's questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Suzanne Kilmer, MD, Principal Investigator — Laser & Skin Surgery Medical Group, Inc.
Locations (1):
- Laser & Skin Surgery Medical Group Inc, Sacramento, California, United States